CLINICAL TRIAL: NCT03491501
Title: Ergonomic Evaluation of Workspaces and Occupational Tasks Targeted for Exoskeleton Support and Definition of Case Studies
Brief Title: Wearable Robotic Upper Body Exoskeleton for Workers
Acronym: Exo4Work
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Prof. Dr., Vrije Universiteit Brussel
Other Study IDs: S000118N
Record Dates: First submitted 2018-03-30; First posted 2018-04-09 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Work-Related Condition; Physical Stress; Mental Fatigue
Keywords: Industrial work; physical effort; mental effort; questionnaires; ergonomic evaluation
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Industrial employees: Ergonomic evaluation using questionnaires in different Industrial settings will be conducted and thus Industrial employees form the included subject group.
  Interventions: Other: Ergonomic evaluation using questionnaires

INTERVENTIONS:
Other: Ergonomic evaluation using questionnaires — Employees will be provided with questionnaires such as the 'Rapid Entire Body Assessment' and NIOSH to obtain information regarding ergonomic working situations

SUMMARY:
The main aim of the project is to evaluate a novel upper body exoskeleton during simulated industrial work. In a first stage of the project, an extensive study involving the end-user companies will be carried out to clearly identify the operator target tasks and typical target task loads for which the exoskeleton will be designed. Based on standard ergonomic evaluation scales (RULA and NIOSH, the Need for Recovery Scale and the Ovako Working Posture Analysing System), high risk tasks will be identified in the field, based on the evaluated information about the workspace configuration, the performed operations and their physical constraints. These will include, but will not be limited to, non-ergonomic postures, for example performing operations above the head or reaching in front, to the side, or behind the body; flexing the arms for extended periods of time; and bending or twisting the torso to lift an object from low or distant locations. Important items to assess in this task are the frequency and duration of tasks and activities, lifting characteristics, perceived physical effort and work-induced fatigue.

ELIGIBILITY:
Inclusion Criteria: Industrial employees

-

Exclusion Criteria:

* non-able bodied individuals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Employees of different companies. Only companies involved in the project will be visited.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-16 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Questionnaire | The time point of data collection: An average of 1yr
  Ergonomic evaluation Industrial work situations

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data of the questionnaires will be shared within the consortium of the project, mainly between sport scientists involved in the project.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data sharing will take place during the experimental process until December 2018.
Access Criteria: Access to data is only possible if partner in the consortium